CLINICAL TRIAL: NCT00610467
Title: Combined MRI and Optical Imaging to Improved Breast Cancer Diagnosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of California, Irvine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Min-Ying (Lydia) Su, Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UCI-HS-2006-5162; R21CA121568 (NIH)
Record Dates: First submitted 2008-01-12; First posted 2008-02-08 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Disease Group (Experimental): Patients with suspicious breast diseases
  Interventions: Device: Disease Group
- Control Group (Experimental): Healthy volunteers for system testing
  Interventions: Device: Control Group

INTERVENTIONS:
Device: Disease Group — Participants will received the following agents before their imaging are taken MRI contrast agent (0.1 mmol/kg) optical contrast agent ICG (0.5 mg/kg)
  Arms: Disease Group
Device: Control Group — Participants will received the following agents before their imaging are taken MRI contrast agent (0.1 mmol/kg) optical contrast agent ICG (0.5 mg/kg)
  Arms: Control Group

SUMMARY:
This study investigates whether adding the optical imaging to magnetic resonance imaging can improve the diagnostic specificity of breast cancer.

DETAILED DESCRIPTION:
This proposal will investigate the performance of a combined optical-MRI imaging system in diagnosis of breast cancer. A diffuse optical tomography (DOT) imaging system will be integrated with a 3.0 T MRI scanner. It is hypothesized that the additional information measured by the combined MRI/DOT system will improve the specificity of DCE-MRI (dynamic contrast enhanced MRI) in diagnosis of breast cancer.

High resolution anatomic MRI and DCE-MRI has evolved into a standard clinical tool for detection and diagnosis of breast lesions. Due to its high sensitivity MRI is fast becoming the most popular imaging modality for screening young women who are susceptible to early development of breast cancer. Pre-operative MRI has also become a common procedure for detecting multifocal or multicentric diseases to facilitate surgical planning. However, despite its high sensitivity, MRI also detects many benign lesions. The low specificity may lead to a great anxiety to patients, and many unnecessary biopsies or over-treatment. Other adjunct imaging modality to improve specificity is greatly needed. MR spectroscopy (MRS) and DOT are two techniques that have great potential to provide complementary information.

After the study is completed, we will be able to test the hypothesis that "additional information provided by MRS and optical imaging can be used in conjunction with morphological and kinetics parameters measured by DCE-MRI to improve diagnostic accuracy of breast cancer". Furthermore, we will be able to determine among these additionally collected information, which parameter(s) are the most essential in improving diagnostic accuracy.

Although the current breast imaging modalities have achieved a high success, further improvements for the subpopulation in whom conventional imaging does not work well are in great need. Our goal is to develop an imaging technology with optimized acquisition protocol to improve diagnosis of breast cancer, particularly for young women with dense breasts who need a breast MRI examination, so that they would not be subjected to false positive findings.

ELIGIBILITY:
Inclusion Criteria:

1. A female older than 21 years of age,
2. Have suspicious imaging findings suggesting a possibility of breast cancer, or biopsy-proven breast cancer.

Exclusion Criteria:

1. Pregnant,
2. Unwilling to give informed consent,
3. Have implanted prosthetic heart valves, pacemaker, neuro-stimulation devices, surgical clips (hemostatic clips) or other metallic implants,
4. Have engaged in occupations or activities which may cause accidental lodging of ferromagnetic materials, or have imbedded metal fragments from military activities,
5. Have received orthodontic work involving ferromagnetic materials,
6. Claustrophobic,
7. Have had allergic response to contrast agents (such as iodine or gadolinium) previously,
8. Have known history of severe renal insufficiency, asthma, allergic conditions, sickle cell anemia, chronic hemolytic anemia, and gastrointestinal disorders.

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2017-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min-Ying Su, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- Center for Functional Onco-Imaging, University of California, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Disease Group | Control Group
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Disease Group | Control Group | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity, Specificity, and Overall Accuracy in Differentiating Between Benign and Malignant Lesions
Description: ROC curves obtained using the regression statistical approach and the artificial neural network will be used to assess the sensitivity, specificity, and overall accuracy in differentiating between benign and malignant lesions. The ROC curves using the optimized morphological and kinetic parameters measured by DCE-MRI will be obtained first, then compared to ROC curves analyzed using the optimized DCE-MRI parameters with the addition of (1) Choline measured by MRS, (2) hemoglobin concentration and oxygen saturation measured by steady state DOT, and (3) transport rates in ICG kinetics measured by dynamic DOT
Time Frame: After we meet the enrollment target
Population: We had performed the combined MRI and optical imaging on two subjects. Due to the small sample size, there is low statistical power to conclude any findings. Study was terminated pre-maturely. All files have been destroyed per IRB requirement. No outcome measure data are available.
Arm/Group | Disease Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Disease group was followed up to 5 years. Healthy volunteer group was monitored for adverse events during imaging visit, and asked about their experiences immediately after imaging and before being released. There were no follow-up period for the healthy volunteer group.
Arm/Group | Disease Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes